CLINICAL TRIAL: NCT00833820
Title: Repetitive Transcranial Magnetic Stimulation in Amyotrophic Lateral Sclerosis
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in Amyotrophic Lateral Sclerosis
Acronym: rTMS-ALS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Vincenzo Di Lazzaro, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 001
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2009-02-02 (Estimated); Status verified 2009-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; transcranial brain stimulation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients receiving real rTMS
  Interventions: Procedure: Real rTMS of the brain
- B (Sham Comparator): patients receiving sham stimulation
  Interventions: Procedure: Sham rTMS of the brain

INTERVENTIONS:
Procedure: Real rTMS of the brain — Repetitive transcranial magnetic stimulation will be performed using a focal coil held over motor cortex on each hemisphere. Stimulation protocol used will be the cTBS in which three pulses of stimulation are given at 50 Hz, repeated every 200 ms for a total of 300 pulses delivered over the right motor cortex. The stimulus intensity will be set at 80% of Action Motor Threshold.
  Arms: A
Procedure: Sham rTMS of the brain — Sham repetitive transcranial magnetic stimulation will be performed using the same stimulator connected to the placebo butterfly coil MCF-P-B-65 which has no stimulating effect on the cortex but produces similar auditory and tactile sensations as the active coil. The site of stimulation and the number of stimuli will be identical to those used for the active magnetic rTMS.
  Arms: B

SUMMARY:
The investigators' preliminary studies demonstrated that repetitive transcranial magnetic stimulation (rTMS) of the brain may determine a slight slowing in the rate of disease progression in ALS patients (Di Lazzaro et al 2004, 2006). The aim of this study is to investigate whether rTMS of the motor cortex performed over a long period of time (12 months) in a group of patients with ALS, can have a more pronounced beneficial effect. The investigators will compare the disease progression in two groups of patients: the first group of patients will be treated with real rTMS (one week daily treatment every month) and the second group of patients will be treated with sham (placebo) rTMS.

DETAILED DESCRIPTION:
Eligible patients should have a diagnosis of definite ALS according to the El Escorial revised criteria with clear clinical upper and lower motor neuron signs. Twenty patients with definite ALS will be enrolled and will be allocated to the treatment: 10 active and 10 sham stimulation. Patients will be randomly allocated by one of the investigators not involved in follow-up evaluations and data analysis. Stratified block randomisation will be performed such that the two treatment groups will be evenly balanced for disease severity, as evaluated with the revised ALS functional rating scale (ALSFRS-R), and duration. The patients and the neurologists assessing the outcomes will be blinded to group assignment.

Outcome measures Patients will be evaluated at the beginning of the treatment and every month until the end of the study at 1 year. At each visit, patients will be evaluated using the ALSFRS-R and manual muscle testing (MMT). MMT testing will be performed by means of the Medical Research Council (MRC) Scale. To obtain an estimate of the overall limb muscle strength we will calculate a MRC compound score by adding the MRC scores of eight upper limb muscles and five lower limb muscles for each side and dividing the sum by the number of muscles tested (26 muscles). We will test the following muscles: biceps brachii, deltoid, triceps brachii, extensor carpi radialis , extensor digitorum communis, abductor digiti minimi, abductor pollicis brevis, opponens pollicis, iliopsoas, rectus femoris, tibialis anterior, extensor hallucis longus, gastrocnemius.

The primary outcome measure will be the rate of decline of ALSFRS-R scores. Secondary outcome measure will be the rate of decline in MMT.

Transcranial brain stimulation Central motor conduction time for the first dorsal interosseous muscle will calculated by subtracting the peripheral conduction time, from spinal cord to muscles, from the latency of responses evoked by cortical stimulation at the maximum stimulator output during voluntary contraction at about 20% of maximum.

Repetitive TMS will be applied over the hand motor area using a MagPro (Medtronic A/S Denmark) stimulator and a figure of eight-shaped coil.

Active rTMS will be performed using the cTBS pattern in which 3 pulses of stimulation are given at 50Hz, repeated every 200 ms for a total of 600 pulses. We will use a butterfly coil (MCF-B-65) with the handle pointed posteriorly and approximately perpendicular to the central sulcus. The initial direction of the current induced in the brain will be posterior-anterior. The stimulation intensity will be 80 % of the active motor threshold (AMT), defined as the minimum single pulse intensity required to produce a motor evoked potential greater than 200 uV on more than five out of ten trials from the contracted contralateral first interosseous muscle. This protocol leads to pronounced and prolonged suppression of cortical excitability that reaches a maximum about 5-10 min after the end of the stimulation.

Sham rTMS will be performed using the same stimulator connected to the placebo butterfly coil MCF-P-B-65 which has no stimulating effect on the cortex but produces similar auditory and tactile sensations as the active coil. The site of stimulation and the number of stimuli will be identical to those used for the active magnetic rTMS.

Repetitive TMS will be performed bilaterally. The order of stimulation of the two hemispheres will be randomized. The stimulation of the two hemispheres will be performed sequentially at an interval of one minute. The motor cortex of each side will be stimulated for five consecutive days every month for twelve consecutive months. In the patients with absent first dorsal interosseous motor evoked potentials after stimulation of one hemisphere, the repetitive stimulation will be performed at the same intensity used for the opposite hemisphere.

Statistical analysis Statistical analysis will be performed using a two-factor (TIME and TREATMENT) repeated measures analysis of variance.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients should have a diagnosis of definite ALS according to the El Escorial revised criteria with clear clinical upper and lower motor neuron signs.

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation:

  * Tracheostomy
  * Pace-maker
  * Implanted metallic devices
  * Epilepsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Rate of decline of ALSFRS-R score | one year

SECONDARY OUTCOMES:
Rate of decline of manual muscle force testing score | one year

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Di Lazzaro, MD, Principal Investigator — Institute of Neurology Università Cattolica Roma
Locations (1):
- Institute of neurology Università Cattolica, Rome, Italy

REFERENCES:
- [Derived] Di Lazzaro V, Pilato F, Profice P, Ranieri F, Musumeci G, Florio L, Beghi E, Frisullo G, Capone F, Sabatelli M, Tonali PA, Dileone M. Motor cortex stimulation for ALS: a double blind placebo-controlled study. Neurosci Lett. 2009 Oct 16;464(1):18-21. doi: 10.1016/j.neulet.2009.08.020. Epub 2009 Aug 12. PMID 19682544